CLINICAL TRIAL: NCT05007262
Title: Clinical Study on the Efficacy and Safety of Tangningtongluo Tablet in Treating Non Proliferative Diabetic Retinopathy - The Syndrome of Yin Asthenia Generating Intrinsic Heat and Eye Collateral Stasis
Brief Title: Tangningtongluo Tablet in the Treatment of Non-proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNTL-21-01
Record Dates: First submitted 2021-08-05; First posted 2021-08-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Type2 Diabetes; Diabetic Retinopathy
Keywords: Diabetes; Retinopathy; Tangningtongluo tablets
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Retinal Diseases | interventions — tangningtongluo; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangningtongluo tablets (Experimental): Tangningtongluo tablets, 4 tablets one time,tid,po, taken after meals.The patients will receive drugs for 24 weeks continuously. After 24 weeks, the researchers will decide whether to continue depend on the patient condition and willingness. The maximum medication time is up to 48 weeks.Basic treatment: According to the comprehensive objectives of China Type 2 Diabetes Guidelines (2020 Edition) .The Angiotensin-Converting Enzyme（ACEI） and Angiotensin Receptor Blocker（ARB） drugs will be continued to use as the original treatment protocol.
  Interventions: Drug: Tangningtongluo tablets
- Calcium dobesilate capsules (Active Comparator): Calcium dobesilate capsules, 1 capsule at a time, tid,po.(morning, midday, and evening), used on an empty stomach.After 24 weeks, the researchers will decide whether to continue depend on the patient condition and willingness. The maximum medication time is up to 48 weeks.Basic treatment: According to the comprehensive objectives of China Type 2 Diabetes Guidelines (2020 Edition) .The Angiotensin-Converting Enzyme（ACEI ）and Angiotensin Receptor Blocker （ARB） drugs will be continued to use as the original treatment protocol.
  Interventions: Drug: Calcium dobesilate capsules

INTERVENTIONS:
Drug: Tangningtongluo tablets — Four pills each time and three times a day after meals.
  Arms: Tangningtongluo tablets
Drug: Calcium dobesilate capsules — 1 capsule at a time, tid,po.(morning, midday, and evening), used on an empty stomach.
  Arms: Calcium dobesilate capsules

SUMMARY:
This trial is planned to collect relevant clinical data to evaluate the prevention efficacy and safety of Tangningtongluo tablets on the non-proliferation period of diabetic retinopathy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks,all patients giving written informed consent will undergo a 1-week screening period to eligibility for study entry.At week 0,patients who meet the eligibility requirements will be randomized into two groups(experimental group and control group)in a 1:1 ratio to Tangningtongluo tablets(4 tablets,tid,po.) or Calcium dobesilate capsules(1 capsule,tid,po.).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with the diagnosis of type 2 diabetes.
* 2. Patients with the diagnosis of non-proliferative diabetic retinopathy and the classified as mild and moderate.
* 3. Target eye best corrected vision acuity (BCVA) ≥ 34 points (ETDRS vision chart, vision equivalent of score 20 / 200, decimal 0.1).
* 4. Patients who meet the syndrome differentiation standards of yin asthenia generating intrinsic heat and eye collateral stasis in traditional Chinese medicine.
* 5. HbA1C ≤ 9%.
* 6. Age between 18 and 75 years old
* 7. Informed consent, voluntary subject. The process of obtaining informed consent form complies with Good Clinical Practice(GCP).

Exclusion Criteria:

* 1. Patient with the diagnosis of diabetic retinopathy is combined with severe vitreous blood effusion, or required total retinal laser treatment or vitrectomy.
* 2. Patient who has been treated with full retinal laser photocoagulation.
* 3. Patient with difficulty in evaluating fundus images with refractive medium turbidity.
* 4. Patient was diagnosed of acute metabolic disorders such as diabetic ketoacidosis or combined with severe acute infection in the past 1 month.
* 5. Patient with other serious diabetes complications, such as diabetes gangrene.
* 6. Patient was allergic to Tangningtongluo tablets, or Calcium dobesilate, or its composition.
* 7. Female patient with pregnancy, or prepare for pregnancy, or lactating.
* 8. Patient with serious cardiovascular, liver, kidney or hematopoietic system disease, and mental diseases.
* 9. Liver and renal function (Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) above 2 x Upper limit of normal (ULN)and Cr> above 1 x Upper limit of normal (ULN)). The diabetic nephropathy stage was 4 and above.
* 10. Patient with eye diseases such as glaucoma, uveitis, optic neuropathy, and severe cataract.
* 11. Patient participated in other clinical researches within a month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Best corrected vision acuity (BCVA) | At 24 weeks
  using ETDRS vision chart measure vision change from Baseline
diabetic retinopathy(DR)progression rate | At 24 weeks
  Using ETDRS Classification to evaluate DR Progress rate

SECONDARY OUTCOMES:
Fundus photography | At 12, 24weeks
  quantitative analysis of fundus microhemangioma, bleeding, exudation, and tube diameter.
Retinal blood oxygen saturation | At 12, 24weeks
  measure retinal blood oxygen saturation
Retinal macular optical coherence tomography angiography (OCTA) | At 12, 24weeks
  measure macular vascular density, retinal thickness, retinal volume;
HbA1c | At 12,24,36 and 48 weeks
  Measure the patient's HbA1c
Routine eye examination; | At 4,8,12, 24,36 and 48 weeks
  Including the examination of cornea, lens, anterior chamber, iris, etc
Efficacy of traditional Chinese medicine syndrome. | At 12, 24 and 48 weeks
  It includes the evaluation of the main symptoms such as blurred vision, dry eyes, secondary symptoms such as mental fatigue, shortness of breath and lazy speech, dry mouth and dry throat and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Junguo Duan, professor, Principal Investigator — Ineye Hospital of Chendu University of TCM
Locations (13):
- China (13):
  - Chongqing hospital of traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital of traditional Chinese Medicine, Lanzhou, Gansu
  - People's Hospital of Anshun City Guizhou Province, Anshun, Guizhou
  - The Second Affiliated Hospital of Guizhou University of traditional Chinese Medicine, Guiyang, Guizhou
  - Hebei Provincial Hospital of traditional Chinese Medicine, Shijiazhuang, Hebei
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Inner Mongolia Hospital of traditional Chinese Medicine, Hohhot, Inner Mongolia
  - Affiliated Hospital of Nantong University, Nantong, Jiangshu
  - Yangzhou Hospital of traditional Chinese Medicine, Yangzhou, Jiangshu
  - Ineye Hospital of Chendu University of TCM, Chengdu, Sichuan
  - Banan Hospital Affiliated to Chongqing Medical University, Chongqing, Sichuan
  - South Central Hospital of Yunnan Province, Honghe Prefecture, Yunnan
  - Eye Hospital of WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No